CLINICAL TRIAL: NCT01803373
Title: A Phase I, Open-label, Randomized, 3-way Crossover Study in 3 Panels of Healthy, Adult Subjects to Assess the Relative Bioavailability of TMC207 Following Single-dose Administration of Two Pediatric Formulations Using a 100 mg Tablet Formulation as the Reference, With and Without Food.
Brief Title: A Study to Assess the Relative Bioavailability of TMC207 Following Single-Dose Administrations of Two Pediatric Formulations in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Infectious Diseases BVBA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR100987; TMC207TBC1002 (Other: Janssen Infectious Diseases BVBA); 2012-005492-13 (EudraCT Number)
Record Dates: First submitted 2013-03-01; First posted 2013-03-04 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2014-03

CONDITIONS: Healthy; Biological Availability
Keywords: Healthy; Biological Availability; Bioavailability; TMC207; Bedaquiline; R207910

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Treatment Sequence ABC (Experimental): Participants in Panel 1 will take the sequence of 3 treatments with a standardized breakfast, participants in Panel 2 will take the sequence of 3 treatments with yogurt, and participants in Panel 3 will take the sequence of 3 treatments after a 10-hour overnight fast (without food). Each treatment in each treatment sequence to be separated by 4 weeks.
  Interventions: Drug: Treatment A (reference); Drug: Treatment B; Drug: Treatment C
- Treatment Sequence ACB (Experimental): Participants in Panel 1 will take the sequence of 3 treatments with a standardized breakfast, participants in Panel 2 will take the sequence of 3 treatments with yogurt, and participants in Panel 3 will take the sequence of 3 treatments after a 10-hour overnight fast (without food). Each treatment in each treatment sequence to be separated by 4 weeks.
  Interventions: Drug: Treatment A (reference); Drug: Treatment B; Drug: Treatment C
- Treatment Sequence BAC (Experimental): Participants in Panel 1 will take the sequence of 3 treatments with a standardized breakfast, participants in Panel 2 will take the sequence of 3 treatments with yogurt, and participants in Panel 3 will take the sequence of 3 treatments after a 10-hour overnight fast (without food). Each treatment in each treatment sequence to be separated by 4 weeks.
  Interventions: Drug: Treatment A (reference); Drug: Treatment B; Drug: Treatment C
- Treatment Sequence BCA (Experimental): Participants in Panel 1 will take the sequence of 3 treatments with a standardized breakfast, participants in Panel 2 will take the sequence of 3 treatments with yogurt, and participants in Panel 3 will take the sequence of 3 treatments after a 10-hour overnight fast (without food). Each treatment in each treatment sequence to be separated by 4 weeks.
  Interventions: Drug: Treatment A (reference); Drug: Treatment B; Drug: Treatment C
- Treatment Sequence CBA (Experimental): Participants in Panel 1 will take the sequence of 3 treatments with a standardized breakfast, participants in Panel 2 will take the sequence of 3 treatments with yogurt, and participants in Panel 3 will take the sequence of 3 treatments after a 10-hour overnight fast (without food). Each treatment in each treatment sequence to be separated by 4 weeks.
  Interventions: Drug: Treatment A (reference); Drug: Treatment B; Drug: Treatment C
- Treatment Sequence CAB (Experimental): Participants in Panel 1 will take the sequence of 3 treatments with a standardized breakfast, participants in Panel 2 will take the sequence of 3 treatments with yogurt, and participants in Panel 3 will take the sequence of 3 treatments after a 10-hour overnight fast (without food). Each treatment in each treatment sequence to be separated by 4 weeks.
  Interventions: Drug: Treatment A (reference); Drug: Treatment B; Drug: Treatment C

INTERVENTIONS:
Drug: Treatment A (reference) — One tablet equivalent to a single 100-mg dose of TMC207 taken orally (by mouth) once.
Drug: Treatment B — Five 20-mg water dispersable tablets equivalent to a single 100-mg dose of TMC207 taken orally (by mouth) once.
Drug: Treatment C — 5 grams (ie,20mg/g) equivalent to a single 100-mg dose of TMC207 taken orally (by mouth) once.

SUMMARY:
The purpose of this study is to test the relative bioavailability (extent and rate to which a drug is taken up by the body) of TMC207 following the administration of two pediatric formulations of TMC207 taken with and without food in healthy adult participants.

DETAILED DESCRIPTION:
This is an open-label (all study staff and participants know the identity of treatments assigned), 3-way cross-over (method used to switch participants from one treatment to another treatment) study. Three panels of 12 healthy adult participants each will be enrolled. Within each panel, participants will be randomly (by chance) assigned to 1 of 6 treatment sequences to receive each of the 3 formulations of TMC207 in a randomized order. The 3 formulations of TMC207 will be referred to as Treatments A, B, and C. In Treatment A, participants will receive a single 100-mg dose of TMC207 formulated as a 100-mg tablet (reference formulation). In Treatment B, participants will receive a single 100-mg dose of TMC207 formulated as 20-mg water dispersible (dissolvable) tablets (i.e. 5 tablets) (pediatric formulation 1). In Treatment C, participants will receive a single 100-mg dose of TMC207 formulated as granules 5 grams (20 mg/g) (pediatric formulation 2). Each treatment will be separated by 4 weeks. Participants in Panel 1 will receive each treatment with a standardized breakfast, Panel 2 will receive each treatment with yogurt, and Panel 3 will receive each treatment after a 10-hour overnight fast (without food). The duration of the treatment period in this study will be 8.5 weeks (includes 4 weeks between treatments).

ELIGIBILITY:
Inclusion Criteria:

* Healthy participant on the basis of physical examination, medical history, vital signs, and electrocardiogram (ECG), and the results of blood biochemistry and hematology tests and a urinalysis performed at screening
* Must have a Body Mass Index (BMI, weight in kg divided by the square of height in meters) of 18.5 to 30.0 kg/m2, extremes included
* Women must be postmenopausal for at least 2 years and have a negative serum pregnancy test at screening and a negative urine pregnancy test at Day -1
* Men must agree to use a highly effective method of birth control (eg., male condom with either female intrauterine device, diaphragm, cervical cap or hormone based contraceptives by their female partner) when having sexual intercourse with a female partner of childbearing potential, and to not donate sperm during the study and for 6 months after receiving the last dose of study drug. Men who have had a vasectomy and have a female partner of childbearing potential must agree to use a male condom during the study and for 6 months after receiving the last dose of study drug
* Participants must be non-smokers for at least 3 months prior to screening

Exclusion Criteria:

* Human immunodeficiency virus - type 1 (HIV-1) or type 2 (HIV-2) infection confirmed at screening
* Hepatitis A, B or C infection confirmed at screening
* A positive urine drug test or alcohol breath test at screening. Urine will be tested for the presence of amphetamines, barbiturates, benzodiazepines, cocaine, methadone, and opioids
* History or any currently active disease or condition that the Investigator considers to be clinically significant for which, in the opinion of the Investigator, participation would not be in the best interest of the participant (eg, compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2013-04; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of TMC207 | Up to 72 hours after study drug intake during 3 treatment sessions
  Protocol-specified pharmacokinetic parameters will be determined from plasma samples collected after each administration of study drug to assess the relative bioavailability of TMC207.

SECONDARY OUTCOMES:
The plasma concentration of the primary metabolite in TMC207 | Up to 72 hours after each study drug intake during 3 treatment sessions
  Protocol-specified pharmacokinetic parameters will be determined from plasma samples collected after each administration of study drug to assess the concentration of the primary metabolite in TMC207.
The effect of food on the relative bioavailability of TMC207 | Up to 72 hours after study drug intake during 3 treatment sessions
  The effect of food will be determined by comparing, across panels, each formulation taken after eating a standardized breakfast versus after eating yoghurt, and versus no food (ie, in the fasted state).
The number of participants reporting adverse events as a measure of safety and tolerability | Up to approximately 12.5 weeks
  Includes up to 30-32 days after the last plasma sample in the last treatment session for participants who complete the study (or up to 30-32 days after a participant withdraws from the study).
The taste of TMC207 | On Day 1 after study drug administration during 3 treatment sessions.
  The taste of each formulation will be assessed by having study participants complete a 5-item questionnaire after they take study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Infectious Diseases BVBA Clinical Trial, Study Director — Janssen Infectious Diseases BVBA
Locations (1):
- Groningen, Netherlands